CLINICAL TRIAL: NCT04505189
Title: Psilocybin as a Treatment for Anorexia Nervosa: A Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19HH5267
Record Dates: First submitted 2020-07-30; First posted 2020-08-10 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psilocybin

STUDY DESIGN:
Masking Description: All participants will receive 3 doses of psilocybin. The maximum dose a participant will receive in a single session is 25 mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin assisted psychotherapy

SUMMARY:
The primary aim of this study is to assess the acceptability and efficacy of treating anorexia nervosa with psilocybin. The secondary aim of this study is to use Magnetic Resonance Imaging (MRI) and Electroencephalography (EEG) to examine the neuronal underpinnings of treatment with psilocybin in this patient group.

DETAILED DESCRIPTION:
Anorexia nervosa is the most fatal of all psychiatric conditions. With the current paucity of effective pharmacological and psychological treatments, and fewer than half of those diagnosed making a full recovery, there is a great need for new treatment avenues to be explored. For this study, we will recruit patients who have a primary diagnosis of anorexia nervosa as defined by DSM-V criteria, which has been established by their specialist ED team to have been present for at least 3 years, and who have found other forms of treatment ineffective. Over a period of 6 weeks, participants who are deemed eligible at screening will partake in 8 study visits, including three psilocybin dosing sessions with varying doses. The maximum dose of psilocybin a participant will receive in a single session is 25 mg. Across these 8 visits, there will also be 2 MRI scans, up to 5 EEG recordings and a range of psychological measures (questionnaires and interviews). There will be a follow-up period of 12 months following the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Primary DSM-V diagnosis of Anorexia Nervosa
2. Current diagnosis of Anorexia Nervosa, established by specialist eating disorder care team to have likely been present for >3 years
3. Current or past treatments have not been successful to maintain remission from anorexia
4. Be in the care of a GP and specialist eating disorder team in the UK
5. Have a GP and specialist eating disorder team in the UK who can confirm diagnosis
6. Sufficiently competent in English and mental capacity to provide written informed consent
7. BMI ≥14kg/m2 and medically stable
8. Capacity to consent
9. Agree to have us maintain contact with an identified next-of-kin for the duration of the study
10. Agree to have us maintain contact with GP and/or specialist eating disorder team as required, for the duration of the study

Exclusion Criteria:

1. Current or previously diagnosed psychotic disorder
2. Immediate family member with a diagnosed psychotic disorder
3. Unstable physical condition e.g., rapid weight loss > 2kg in the prior month
4. Abnormal serum electrolytes, raised cardiac enzymes, hepatic or renal dysfunction
5. MRI or EEG contraindications
6. A history of laxative abuse in the last 3 months (more than twice a week for 3 months)
7. History of serious suicide attempts or presence of a suicide/ serious self-harm risk at screening
8. Currently an involuntary patient
9. Emotionally unstable personality, history of mania, or other psychiatric problem that the screening clinician feels may jeopardise the therapeutic alliance and/or safe exposure to psilocybin
10. Blood or needle phobia
11. Positive pregnancy test at screening or during the study, or woman who are breastfeeding
12. If sexually active, participants who lack appropriate contraceptive measures
13. Drug or alcohol dependence within the last 6 months
14. No email access
15. Patients presenting with abnormal QT interval prolongation at screening or with a history of this (QTc at screening above 470ms)
16. Patients who are currently, or have recently (within 3 months) been enrolled in another CTIMP.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Readiness and Motivation Questionnaire (RMQ) | Baseline - Primary endpoint (6 weeks)
  Increase in readiness and motivation to recover from baseline to primary endpoint, which will be related to long-term improvements in psychopathology.
Eating Disorder Examination (EDE) | Baseline - Primary endpoint (6 weeks) - 6 month follow-up.
  Decrease in eating disorder psychopathology.
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline - Primary endpoint (6 weeks) - 6 month follow-up.
  Decrease in eating disorder psychopathology.

SECONDARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) | Baseline - Primary endpoint (6 weeks)
  Changes in blood oxygen level dependent (BOLD) signal during rest and disorder relevant tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Hammersmith campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spriggs MJ, Douglass HM, Park RJ, Read T, Danby JL, de Magalhaes FJC, Alderton KL, Williams TM, Blemings A, Lafrance A, Nicholls DE, Erritzoe D, Nutt DJ, Carhart-Harris RL. Study Protocol for "Psilocybin as a Treatment for Anorexia Nervosa: A Pilot Study". Front Psychiatry. 2021 Oct 20;12:735523. doi: 10.3389/fpsyt.2021.735523. eCollection 2021. PMID 34744825